CLINICAL TRIAL: NCT04466826
Title: Transnasal Sphenopalatine Ganglia Block for Management of Chronic Migraines in Pediatric Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202006033
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Migraine in Children; Pain, Neuropathic
MeSH Terms: conditions — Neuralgia | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Intervention Model Description: Open label, pre/post-treatment pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Minors with chronic migraines (Experimental)
  Interventions: Other: Headache Journal; Drug: Sphenopalatine Block; Device: Tx360

INTERVENTIONS:
Other: Headache Journal — Phase 1 of study to determine a baseline for headache frequency, headache intensity and medication usage patterns
Drug: Sphenopalatine Block — Phase 2 of study providing medication using 0.3ml of 0.5% Bupivacaine per nares delivered intranasal via the Tx360 device
Device: Tx360 — Phase 2 of study providing medication using 0.3ml of 0.5% Bupivacaine per nares delivered intranasal via the Tx360 device

SUMMARY:
Single-center, open-label, pre-post treatment pilot study to evaluate the safety and effectiveness of sphenopalatine ganglia blocks for the treatment of chronic migraine in the pediatric population. 50 children with a diagnosis of chronic migraines will undergo a series of three transnasal sphenopalatine ganglia blocks to measure their effect on headache frequency, headache intensity, headache duration, and use of headache medication.

ELIGIBILITY:
Inclusion Criteria:

Children ages 8 to 17 years old Meet the criteria for chronic migraines Have remained stable on their current headache medication for a minimum of 4 weeks.

Able to provide informed consent from parent or legal guardian Able to provide assent if subject is a minor of appropriate age

Exclusion Criteria:

Allergy to local anesthetic Developmental delay (e.g. non-verbal) Inability to use numeric pain scale Inability to perform or tolerate transnasal procedure Substance abuse disorders Known pregnancy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Reduction in frequency of headache days: pre-treatment | Up to 4 weeks following consent
  Weekly headache journal check in - 5 questions with y/n answers and free text entry
Reduction in frequency of headache days: post-treatment | Up to one year following consent
  Weekly headache journal check in - 5 questions with y/n answers and free text entry

SECONDARY OUTCOMES:
Maximum headache severity: pre-treatment | up to 4 weeks following consent
  Participant records headache intensity on headache journal. Scale is 0-10, with 0 being the least severity and 10 being the worst severity
Maximum headache severity: post-treatment | up to one year following consent
  Participant records headache intensity on headache journal. Scale is 0-10, with 0 being the least severity and 10 being the worst severity
Headache duration: pre-treatment | Up to 4 weeks following consent
  Participant records headache duration by documenting the start and end time of the headache
Headache duration: post-treatment | Up to one year following consent
  Participant records headache duration by documenting the start and end time of the headache
Use of rescue medication: pre-treatment | Up to 4 weeks following consent
  Participant records use with a y/n answer and provides the name of the medication
Use of rescue medication: post-treatment | Up to one year following consent
  Participant records use with a y/n answer and provides the name of the medication

CONTACTS AND LOCATIONS:
Overall Officials: Jacob AuBuchon, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Abu-Arafeh I, Razak S, Sivaraman B, Graham C. Prevalence of headache and migraine in children and adolescents: a systematic review of population-based studies. Dev Med Child Neurol. 2010 Dec;52(12):1088-97. doi: 10.1111/j.1469-8749.2010.03793.x. Epub 2010 Sep 28. PMID 20875042
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Wober-Bingol C. Epidemiology of migraine and headache in children and adolescents. Curr Pain Headache Rep. 2013 Jun;17(6):341. doi: 10.1007/s11916-013-0341-z. PMID 23700075